CLINICAL TRIAL: NCT04683107
Title: Efficacy of Eccentric Versus Isometric Exercise in Reducing Pain in Runners With Proximal Hamstring Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Haifa (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: University of Haifa (UHaifa)
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Proximal Hamstring Tendinopathy; Tendinopathy; Eccentric Exercise; Isometric Exercise; Hamstring Tendon Injury
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric protocol (Experimental)
  Interventions: Other: Eccentric protocol
- Isometric protocol (Experimental)
  Interventions: Other: Isometric protocol

INTERVENTIONS:
Other: Eccentric protocol — Participants in this arm will perform progressive eccentric exercise protocol
  Arms: Eccentric protocol
Other: Isometric protocol — Participants in this arm will perform progressive isometric exercise protocol
  Arms: Isometric protocol

SUMMARY:
Tendon injuries are the most common injuries in sports. They are difficult to treat and cause prolonged absence and decreased athlete performance. Proximal hamstring tendinopathy (PHT) is one of them. First described by Puranen and Orava in 1988 as hamstring syndrome. This injury is most common in the active population.

PHT is a chronic degenerative injury that is produced by mechanical overload and repetitive stretch. Risk factors include overuse, poor lumbopelvic stability and relative weakness of the hamstring muscles. The phenomenon manifests itself with deep pain in the ischial tuberosity area and projection to the posterior thigh, pain during prolonged sitting, pain during hip flexion and knee extension and pain that increases or arises during running, especially during the swing phase.

Risk factors are divided into internal (systemic and biomechanical) and external factors. Internal factors associated with systemic characteristics, include advanced age, sex, obesity, genetics, inflammation and autoimmune conditions, diabetes, hyperlipidemia, and drug use. The external factors, which are more modifiable, are those that depend on the patient's external environment and include training errors such as increasing training volume and / or intensity too quickly and insufficient recovery that cause an overload on the tendon.

For PHT two conditions are considered provocative - energy storage, an action that is typical in the late swing phase while running and repetitive movements that cause compressive forces of the tendon on ischial tuberosity. Compressive forces increase as the hip or trunk flex which explains why training errors such as an increase in volume or intensity of the training and non-gradual change in training type, such as hurdle or hills training, are considered to be factors involved in PHT.

PHT treatment options include physiotherapy, shock waves, Platelet rich plasma (PRP) and surgical treatment. Non-surgical treatments for tendinopathy includes gradual loading of the tendon under the supervision of the level of pain. The load on the tendon causes an increase in collagen synthesis and an increase in the stiffness and capacity of the tendon which ultimately helps return the athlete to function and reduces the level of pain.

Although the injury mechanism is common among runners and athletes from various endurance disciplines (medium and long distance runners, triathletes, etc.) the phenomenon and its treatment has not been sufficiently studied within this population.

ELIGIBILITY:
Inclusion Criteria:

* Medium and long distance runners and endurance athletes (triathlon, Iron Man)
* over the age of 40
* With tendon pain lasting 3 months or more, at the location of hamstring insertion in Ischial tuberosity, that increases during or after running.

Exclusion Criteria:

* Hamstring tear (posterior thigh muscle) according to MRI
* Stress fractures of the ischium bone
* Radiated pain in the posterior thigh originating in the lumbar spine, hip joint or sacroiliac joint
* Other pathologies or rupture of the hamstring muscle
* Exclude people who have received therapeutic intervention in the last month
* Medication use for PHT
* Pain located medially or laterally to the Ischial tuberosity
* Pregnant women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Victorian Institute of Sport Assessment-Proximal Hamstring Tendons (VISA-H) questionnaire | 6 weeks
  VISA-H is a patient reported outcome questionnaire with high psychometric properties for measuring pain, function and sporting activity in patients with PHT
Isometric and eccentric muscle force | 6 weeks
Running performance | 6 weeks
  measuring running time for 1.5 km